CLINICAL TRIAL: NCT02121093
Title: Effect of Vibration Stimulation Applied to Different Frequencies in Cortical Excitability and Muscular Function: Randomised Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade do Vale do Paraíba (Other)
Responsible Party: Principal Investigator, Izabela dos Santos Mendes, Effect of vibration stimulation applied to different frequencies in cortical excitability and muscular function: randomised clinical trial, Universidade do Vale do Paraíba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: janaina de moraes silva
Record Dates: First submitted 2014-04-07; First posted 2014-04-23 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Healthy
Keywords: vibration; physiotherapy; cortex; muscles
MeSH Terms: interventions — Vibration

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- alpha band of the EEG and electromyographic activity (No Intervention): - 20 will be in the evaluation group (EG); then review the alpha band of EEG and EMG activity.
- Vibration (Experimental): * • 20 vai participar no grupo de baixa freqüência de vibração estimulação (LFVS);
  * 20 no grupo de estimulação da vibração de média freqüência (MFVS);
  * 20 vai participar no grupo de alta freqüência de vibração estimulação (HFVS). then review the alpha band of EEG and EMG activity.
  Interventions: Procedure: vibration

INTERVENTIONS:
Procedure: vibration
  Arms: Vibration

SUMMARY:
The vibration stimulation is regarded as a new method of training and therapy to change afferent parts and cortical projections, which are important for motor control. This study aims to check effects of different frequency parameters for electrical cortical potentials and electrical muscular potentials in healthy young adults. 80 volunteers will participate in the study, and they will be randomly subdivided in four groups for trials. The methodology consists of electroencephalographic and electromyographic assessment before and after 15-minute vibration application with a digital vibratory pad.

DETAILED DESCRIPTION:
The vibratory stimulation is regarded as a new training method and capable of modulating peripheral afferents and cortical projections therapy, which are important in motor control. This study aims to determine the effects of different parameters on cortical frequency electric potential and electric potential muscle in healthy young adults. Will participate in the study 80 volunteers, these randomly divided into four groups for the experimental procedures. The methodological approach consists of an electroencephalographic and electromyographic evaluation before and after 15 minutes of application of vibration through a digital vibrating pad.

ELIGIBILITY:
Inclusion Criteria:

* Physically and mentally healthy
* Right-handed volunteers who are not using psychoactive or psychotropic substances,
* Have nourished themselves up to three hours before the experiment.

Exclusion Criteria:

* Under 18-year- and over-60-old volunteers
* who do not fit into using data collection equipment,
* individuals who have slept less than six to eight hours the night before the experiment,
* who have already undergone vibration training and had problems with using it.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-05; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Effect of vibration stimulation applied to different frequencies in cortical excitability and muscular function: randomised clinical trial | 1 month
  We know that the vibration has multiple physiologic effects, promoting normal patterns of motor activity by changing motor-neuron excitability. Vibrations increase the final afferent influx of the primary muscular fuse, allowing the reflex contraction, the so-called tonic vibration reflex . This reflex is mediated by both segmental and supra-segmental spine path, and is supported by upper centres.
Effect of vibration stimulation applied to different frequencies in cortical excitability and muscular function: randomised clinical trial | 1 month
  The 80 volunteers will be randomly gathered in study groups by random computer-given numbers.
  From these 80 volunteers, 20 will be in the evaluation group (EG); 20 will participate in the group of low-frequency vibration stimulation (LFVS); 20 in the group of medium-frequency vibration stimulation (MFVS); and 20 will take part in the group of high-frequency vibration stimulation (HFVS).
Effect of vibration stimulation applied to different frequencies in cortical excitability and muscular function: randomised clinical trial | 1 month
  The 80 volunteers will be randomly gathered in study groups by random computer-given numbers.
  From these 80 volunteers, 20 will be in the evaluation group (EG); 20 will participate in the group of low-frequency vibration stimulation (LFVS); 20 in the group of medium-frequency vibration stimulation (MFVS); and 20 will take part in the group of high-frequency vibration stimulation (HFVS).
  The three groups is intended to observe increased alpha band

SECONDARY OUTCOMES:
Effect of vibration stimulation applied to different frequencies in cortical excitability and muscular function: randomised clinical trial | 1 month
  The 80 volunteers will be randomly gathered in study groups by random computer-given numbers.
  From these 80 volunteers, 20 will be in the evaluation group (EG); 20 will participate in the group of low-frequency vibration stimulation (LFVS); 20 in the group of medium-frequency vibration stimulation (MFVS); and 20 will take part in the group of high-frequency vibration stimulation (HFVS).
  The three groups is intended to observe increased electromyographic activity of the muscles

CONTACTS AND LOCATIONS:
Locations (1):
- Janaina de Moraes Silva, Teresina, Piauí, Brazil